



# Official Title of Study:

A Randomized Control Trial Examining the Treatment Efficacy of a Novel Approach to Cognitive Remediation in Public Safety Personnel with Post-Traumatic Stress Disorder (PTSD) and Co-morbid Conditions

Date of Document:

August 9, 2019

**Document Uploaded:** 

August 21, 2019





## Dear Potential Participant,

You are invited to participate in the **Goal Management Therapy** project conducted by Dr. Margaret McKinnon, PhD, C.Psych. at Homewood Research Institute, in Guelph, ON. This study aims to examine if a cognitive training program called Goal Management Therapy (GMT) is effective in reducing cognitive difficulties, and improving every-day functioning in Public Safety Personnel and Military/Veterans with post-traumatic stress disorder (PTSD).

Participation in this study is voluntary. In order to determine whether or not you want to take part in this research study, you should understand what is involved and the potential risks and benefits. Please take your time to review this letter of information. You may discuss it with your friends, family, or members of your clinical care team before making your decision.

### Why is this research being done?

Research has shown that individuals with PTSD often experience difficulties in many parts of cognitive functioning, like memory, learning, and attention. Such difficulties can have negative impacts, including less productivity at work or home and changes in social functioning. At present, very little research has been done to investigate whether cognitive difficulties can be targeted through a specific treatment approach. In this study, we plan to investigate the effectiveness of an approach known as Goal Management Therapy (GMT) in reducing cognitive difficulties and improving day-to-day functioning (i.e., work or social functioning) in individuals with PTSD. We are also interested in whether GMT is more effective than the standard treatment for cognitive difficulties in PTSD: psychosocial education. For this reason, participants will be randomly assigned to either a GMT group or a psychosocial education group. Should this study be successful, it has the potential to have a positive impact on people with these disorders, their families, and society. Specifically, if we demonstrate that GMT can reduce difficulties in cognitive functioning and improve day-to-day functioning in the study group, we can expect that it would also be successful for others with PTSD.

## What are the possible risks and discomforts?

Your participation in this study will include disclosure of personal information regarding your symptoms and difficulties related to PTSD, and your history of exposure to traumatic events. This may cause you to feel embarrassed, uncomfortable, or become distressed. You are not required to answer any questions if you do not wish to and the research team will make every effort to minimize these risks.

### **How to Participate:**

If you are interested in receiving more information, please fill out the contact form. A research team member will contact you to see if you are eligible to participate. Completing the contact form does **not** mean you have given consent to participate.





## **Questions:**

If you have any questions about the study, please contact Dr. Margaret McKinnon at 519-824-1010 ext. 32498. If you have any questions regarding your rights as a research participant, you may contact Dr. Steve Abdool, Bioethicist & Director, Regional Centre for Excellence in Ethics, Homewood Health Centre at SAbdool@homewoodhealth.com or (519) 824-1010 Ext. 32118.





#### **Consent to Contact**

My signature on this consent form means:

- I agree that Homewood Research Institute (HRI) can contact me using the telephone number or email address provided to inquire about participating in the Goal Management Therapy research project.
- I understand that my signature below does not mean I am a participant in the project
- I understand if I do not want to be contacted anymore I can let HRI know by contacting 519-824-1010 ext. 32180 or <a href="https://example.com"><u>HMillman@Homewoodhealth.com</u></a>

| Participant's name (please print): | Researcher's name (please print): |
|---|---|
| Participant's Signature: | Researcher's Signature: |
| Date: | Date: |
| Con Please print clearly. | tact Information |
| First Name: | Last Name: |
| Telephone Number: | |
| Email Address: | |
| City: | |
| What is your preferred method of contact Phone Email Either | t? |
| What is your preferred time to be contact | ed by phone? |
| Morning (9am-12pm) Afternoo | n (12pm-4pm) Evening (4pm-8pm) |
| Anytime (9am-8pm) | |